CLINICAL TRIAL: NCT03828747
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy, and Safety Study of MTAU9937A in Patients With Moderate Alzheimer's Disease
Brief Title: A Study of Semorinemab in Patients With Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GN40040
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Results first posted 2022-10-03 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — (18F)GTP1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semorinemab (Experimental): Semorinemab will be administered intravenously in the double-blind treatment period, and semorinemab will be administered intravenously in the optional open-label extension period.
  Interventions: Drug: Semorinemab; Drug: [18F]GTP1
- Placebo (Placebo Comparator): Placebo will be administered intravenously in the double-blind treatment period and semorinemab will be administered intravenously in the optional open-label extension.
  Interventions: Drug: Placebo; Drug: [18F]GTP1

INTERVENTIONS:
Drug: Semorinemab — Participants will receive semorinemab every 2 weeks (Q2W) for the first three doses of the double-blind treatment period and every 4 weeks (Q4W) thereafter during the double-blind treatment period. Semorinemab will be administered Q4W in the OLE period.
  Other Names: MTAU9937A; RO7105705
  Arms: Semorinemab
Drug: Placebo — Participants will receive placebo every 2 weeks (Q2W) for the first three doses of the double-blind treatment period and every 4 weeks (Q4W) thereafter during the double-blind treatment period.
  Arms: Placebo
Drug: [18F]GTP1 — [18F]GTP1 will be administered as a solution for intravenous (IV) use, as part of positron emission tomography (PET) imaging.

SUMMARY:
This Phase II, multicenter, randomized, double-blind, placebo-controlled, parallel-group study will evaluate the clinical efficacy, safety, pharmacokinetics, and pharmacodynamics of semorinemab in patients with moderate AD. The study consists of a screening period, a double-blind treatment period, an optional open-label extension (OLE) period, and a safety follow-up period. There may be up to two study cohorts.

ELIGIBILITY:
Inclusion Criteria:

* National Institute on Aging/Alzheimer's Association core clinical criteria for probable AD dementia
* Evidence of the AD pathological process, by a positive amyloid assessment either on CSF Aβ1-42 as measured on Elecsys β-Amyloid(1-42) Test System OR amyloid PET scan
* AD dementia of moderate severity, as defined by a screening MMSE score of 16-21 points, inclusive, and a CDR-GS of 1 or 2
* Availability of a person with sufficient contact with the participant to be able to provide accurate information on the participant's cognitive, behavioral and functional ability

Exclusion Criteria:

* Pregnant or breastfeeding
* Inability to tolerate MRI procedures or contraindication to MRI
* Contraindication to PET imaging
* Residence in a skilled nursing facility
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study, or bias the assessment of the clinical or mental status of the participant to a significant degree
* Any evidence of a condition other than AD that may affect cognition
* Substance abuse within the past 2 years
* Use of any experimental therapy within 90 days or 5 half-lives prior to screening, whichever is greater, or any passive immunotherapy against tau
* Use of any passive immunotherapy (immunoglobulin) against Aβ, unless the last dose was at least 1 year prior to screening or any active immunotherapy (vaccine) that is under evaluation to prevent or postpone cognitive decline
* Any other biologic therapy or previous treatment with medications specifically intended to treat Parkinsonian symptoms or any other non-AD neurodegenerative disorder within 1 year of screening
* Systemic immunosuppressive therapy within 12 months of screening through the entire study period
* Typical antipsychotic or neuroleptic medication within 6 months of screening
* Daily treatment with any of the following classes of medication (except for intermittent short-term use): opiates or opioids, benzodiazepines, barbiturates, hypnotics, or any medication with clinically significant centrally-acting antihistamine or anticholinergic activity
* Stimulant medications, unless the dose has been stable within the 6 months prior to screening and is expected to be stable throughout the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (49):
- United States (31):
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Stanford University; Stanford Clinical Cancer Ctr, Palo Alto, California
  - Pacific Research Network - PRN, San Diego, California
  - Molecular Neuroimaging; MRI/PET, New Haven, Connecticut
  - KI Health Partners, LLC; New England Institute for Clinical Research, Stamford, Connecticut
  - JEM Research LLC, Atlantis, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Neuropsychiatric Research; Center of Southwest Florida, Fort Myers, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Synexus Clinical Research US, Inc. - Orlando, Orlando, Florida
  - Alzheimer?s Research and Treatment Center, Wellington, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Rush University Medical Center - Chicago, Chicago, Illinois
  - Alexian Brothers Neuroscience Institute, Elk Grove Village, Illinois
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - Brigham and Womens Hospital; Center for Alzheimer Research & Treatment, Boston, Massachusetts
  - Alzheimers Disease Center, Quincy, Massachusetts
  - Center for Memory and Aging, Saint Paul, Minnesota
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Empire Neurology PC; MS Center of Northeastern NY, Latham, New York
  - University of Rochester; AD-CARE, Rochester, New York
  - Summit Research Network Inc., Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital; Movement Disorders Program, Providence, Rhode Island
  - Neurology Clinic PC, Cordova, Tennessee
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - The Memory Clinic, Bennington, Vermont
- France (5):
  - Chu Toulouse, Bron
  - CHU de la Timone - Hopital d Adultes; Service de Neurologie, Marseille
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - Hopital des Charpennes, Villeurbanne
- Poland (7):
  - Podlaskie Centrum Psychogeriatrii, Bia?ystok
  - Novo-Med Zielinski i wspolnicy Sp. j., Katowice
  - NZOZ NEURO-KARD Ilkowski i Partnerzy Sp. Partn. Lek, Późna
  - Osrodek Badan Klinicznych Euromedis, Szczecin
  - Centrum Medyczne NeuroProtect, Warsaw
  - Centrum Medyczne AMED, Warsaw
  - NZOZ WCA, Wroc?aw
- Spain (6):
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Fundacio ACE, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neurologia, Barcelona
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm)

REFERENCES:
- [Derived] Chandler JM, Lansdall CJ, Ye W, McDougall F, Belger M, Toth B, Mi X, Sink KM, Atkins AS. The Alzheimer's Disease Cooperative Study - Activities of Daily Living dependence score: revision and validation of an algorithm evaluating patient dependence across the spectrum of AD severity. J Prev Alzheimers Dis. 2025 Sep;12(8):100261. doi: 10.1016/j.tjpad.2025.100261. Epub 2025 Jul 1. PMID 40603145
- [Derived] Schauer SP, Toth B, Lee J, Honigberg LA, Ramakrishnan V, Jiang J, Kollmorgen G, Bayfield A, Wild N, Hoffman J, Ceniceros R, Dolton M, Bohorquez SMS, Hoogenraad CC, Wildsmith KR, Teng E, Monteiro C, Anania V, Yeh FL. Pharmacodynamic effects of semorinemab on plasma and CSF biomarkers of Alzheimer's disease pathophysiology. Alzheimers Dement. 2024 Dec;20(12):8855-8866. doi: 10.1002/alz.14346. Epub 2024 Nov 8. PMID 39513754
- [Derived] Monteiro C, Toth B, Brunstein F, Bobbala A, Datta S, Ceniceros R, Sanabria Bohorquez SM, Anania VG, Wildsmith KR, Schauer SP, Lee J, Dolton MJ, Ramakrishnan V, Abramzon D, Teng E; Lauriet investigators. Randomized Phase II Study of the Safety and Efficacy of Semorinemab in Participants With Mild-to-Moderate Alzheimer Disease: Lauriet. Neurology. 2023 Oct 3;101(14):e1391-e1401. doi: 10.1212/WNL.0000000000207663. Epub 2023 Aug 29. PMID 37643887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 49 centers in 4 countries.
Pre-assignment Details: A total of 272 participants were enrolled at 49 centers.
Groups:
- Semorinemab: Semorinemab was administered intravenously in the double-blind treatment period and was administered intravenously in the optional open-label extension period.
- Placebo: Placebo was administered intravenously in the double-blind treatment period and semorinemab was administered intravenously in the optional open-label extension.
Period: Double-Blind Treatment Period
Arm/Group | Semorinemab | Placebo
Started | 136 | 136
Cohort 1 (Participants who completed the double-blind treatment period (before implementation of Protocol Version 3), or participants who completed the double-blind study drug treatment through Week 45 without any missed doses of study drug (after implementation of Protocol Version 4), were assigned to Cohort 1. In Cohort 1, the double-blind treatment period has a duration of 48 weeks.) | 92 | 99
Cohort 2 (Participants who were active in the double-blind treatment period (after implementation of Protocol Version 3) or participants who missed one or more study drug dose (after implementation of Protocol version 4) were assigned to Cohort 2. In Cohort 2, the double-blind treatment period has a duration of 60 weeks.) | 43 | 33
Completed | 106 | 102
Not Completed | 30 | 34
Not completed — Adverse Event | 6 | 6
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 17 | 19
Not completed — Physician Decision | 1 | 4
Not completed — Various reasons | 5 | 3
Period: Open-Label Extension
Arm/Group | Semorinemab | Placebo
Started | 102 | 97
Completed | 48 | 52
Not Completed | 54 | 45
Not completed — Adverse Event | 9 | 7
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 31 | 30
Not completed — Various reasons | 4 | 4
Not completed — Physician Decision | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semorinemab | Placebo | Total
Number analyzed (Participants) | 136 | 136 | 272
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.6 (8.2) | 73.0 (8.0) | 72.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 84 | 176
  Male | 44 | 52 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 117 | 115 | 232
  Unknown or Not Reported | 15 | 18 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 122 | 119 | 241
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Last Visit of Double-Blind Treatment Period in Cognitive Function as Measured by the Alzheimer's Disease Assessment Scale, Cognitive Subscale, 11-Item Version (ADAS-Cog11)
Description: The Alzheimer's Disease Assessment Scale, Cognitive Subscale, 11-Item Version (ADAS-Cog11) is an 11 item cognitive subscale used to quantify the areas of cognitive function most often affected in Alzheimer's disease. The total score ranges from 0-70 with lower scores indicating better cognitive function.
Time Frame: Baseline to Week 49 for Cohorts 1 and 2, and Baseline to Week 61 for Cohort 2
Population: The modified intent-to-treat population included all randomized participants who received at least one dose of study drug and had at least one baseline and one postbaseline ADAS-Cog11 score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 123 | 115
Units on a scale
  Baseline | 23.93 (0.533) | 24.09 (0.589)
  Change from Baseline at Week 49 (includes Cohort 1 and 2): number analyzed (Participants) | 102 | 96
  Change from Baseline at Week 49 (includes Cohort 1 and 2) | 3.96 (0.658) | 6.85 (0.643)
  Change from Baseline at Week 61 (only Cohort 2): number analyzed (Participants) | 38 | 30
  Change from Baseline at Week 61 (only Cohort 2) | 5.71 (0.907) | 8.47 (0.965)
Statistical Analysis 1: Comparison: Semorinemab vs Placebo; Change from Baseline at Week 49; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Least Squares Mean Difference = -2.89, 95% CI 2-sided [-4.56 to -1.21], Standard Error of Mean 0.849
Statistical Analysis 2: Comparison: Semorinemab vs Placebo; Change from Baseline at Week 61; Test type: Superiority; p = 0.0351, Mixed Models Analysis; Least Squares Mean Difference = -2.75, 95% CI 2-sided [-5.31 to -0.20], Standard Error of Mean 1.287

2. Primary Outcome: Change From Baseline to Last Visit of Double-Blind Treatment Period in Functional Capacities as Measured by the Alzheimer's Disease Cooperative Study-Daily Living Inventory (ADCS-ADL)
Description: The Alzheimer's Disease Cooperative Study-Daily Living Inventory (ADCS-ADL) is a scale used to quantify performance of activities of daily living (ADL). Scores on the ADCS-ADL range from 0-78, with higher scores indicating better ADL function.
Time Frame: Baseline to Week 49 for Cohorts 1 and 2, and Baseline to Week 61 for Cohort 2
Population: The modified intent-to-treat population included all randomized participants who received at least one dose of study drug and had at least one baseline and one postbaseline ADAS-Cog11 and the ADCS-ADL score at the given time point.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 123 | 115
Units on a scale
  Baseline | 62.03 (0.764) | 59.74 (0.842)
  Change from Baseline at Week 49 (includes Cohort 1 and 2): number analyzed (Participants) | 107 | 101
  Change from Baseline at Week 49 (includes Cohort 1 and 2) | -7.63 (1.002) | -6.80 (0.974)
  Change from Baseline at Week 61 (only Cohort 2): number analyzed (Participants) | 40 | 33
  Change from Baseline at Week 61 (only Cohort 2) | -9.29 (1.343) | -7.57 (1.462)
Statistical Analysis 1: Comparison: Semorinemab vs Placebo; Change from Baseline at Week 49; Test type: Superiority; p = 0.5207, Mixed Models Analysis; Least Squares Mean Difference = -0.83, 95% CI [-3.39 to 1.72], Standard Error of Mean 1.295
Statistical Analysis 2: Comparison: Semorinemab vs Placebo; Change from Baseline at Week 61; Test type: Superiority; p = 0.3704, Mixed Models Analysis; Least Squares Mean Difference = -1.72, 95% CI [-5.50 to 2.07], Standard Error of Mean 1.911

3. Secondary Outcome: Change From Baseline to Last Visit of Double-Blind Treatment Period on the Clinical Dementia Rating-Sum of Boxes (CDR-SB)
Description: The Clinical Dementia Rating-Sum of Boxes (CDR-SB) is a scale used to quantify the severity of symptoms of dementia. The CDR-SB is obtained through interviews of patients and informants, and disease severity is rated in 6 domains of functioning: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a 5-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). The CDR-SB score is obtained by summing each of the domain box scores, with scores ranging from 0 to 18, with the higher values representing more severe impairment.
Time Frame: Baseline to Week 49 for Cohorts 1 and 2, and Baseline to Week 61 for Cohort 2
Population: The modified intent-to-treat population included all randomized participants who received at least one dose of study drug and had at least one baseline and one postbaseline ADAS-Cog11 and the CDR-SB score at the given time point.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 123 | 115
Units on a scale
  Baseline | 6.23 (0.156) | 6.51 (0.182)
  Change from Baseline at Week 49 (includes Cohort 1 and 2): number analyzed (Participants) | 109 | 101
  Change from Baseline at Week 49 (includes Cohort 1 and 2) | 1.80 (0.217) | 1.54 (0.214)
  Change from Baseline at Week 61 (only Cohort 2): number analyzed (Participants) | 40 | 33
  Change from Baseline at Week 61 (only Cohort 2) | 2.45 (0.367) | 2.28 (0.393)
Statistical Analysis 1: Comparison: Semorinemab vs Placebo; Change from Baseline at Week 49; Test type: Superiority; p = 0.3501, Mixed Models Analysis; Least Squares Mean Difference = 0.26, 95% CI [-0.29 to 0.82], Standard Error of Mean 0.282
Statistical Analysis 2: Comparison: Semorinemab vs Placebo; Change from Baseline at Week 61; Test type: Superiority; p = 0.7431, Mixed Models Analysis; Least Squares Mean Difference = 0.17, 95% CI 2-sided [-0.87 to 1.22], Standard Error of Mean 0.525

4. Secondary Outcome: Change From Baseline to Last Visit of Double-Blind Treatment Period on the Mini-Mental State Examination (MMSE)
Description: The Mini Mental State Examination (MMSE) is a brief clinical cognitive examination commonly used to screen for dementia and other cognitive deficits that has a total score of 0-30. Higher scores indicate better cognitive function.
Time Frame: Baseline to Week 49 for Cohorts 1 and 2, and Baseline to Week 61 for Cohort 2
Population: The modified intent-to-treat population included all randomized participants who received at least one dose of study drug and had at least one baseline and one postbaseline ADAS-Cog11 and the MMSE score at the given time point.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 123 | 115
Units on a scale
  Baseline | 18.38 (0.182) | 18.15 (0.197)
  Change from Baseline at Week 49 (includes Cohort 1 and 2): number analyzed (Participants) | 105 | 97
  Change from Baseline at Week 49 (includes Cohort 1 and 2) | -2.86 (0.330) | -3.12 (0.325)
  Change from Baseline at Week 61 (only Cohort 2): number analyzed (Participants) | 39 | 29
  Change from Baseline at Week 61 (only Cohort 2) | -3.14 (0.429) | -4.22 (0.466)
Statistical Analysis 1: Comparison: Semorinemab vs Placebo; Change from Baseline at Week 49; Test type: Superiority; p = 0.5366, Mixed Models Analysis; Least Squares Mean Difference = 0.27, 95% CI [-0.58 to 1.11], Standard Error of Mean 0.429
Statistical Analysis 2: Comparison: Semorinemab vs Placebo; Change from Baseline at Week 61; Test type: Superiority; p = 0.0851, Mixed Models Analysis; Least Squares Mean Difference = 1.08, 95% CI [-0.15 to 2.30], Standard Error of Mean 0.618

5. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An Adverse Event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to end of study (approximately 4 years and 7 months)
Population: The safety population included all randomized participants who received at least one dose of either semorinemab or placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Semorinemab (Open-label Extension): Semorinemab was administered intravenously in the optional open-label extension period.
Arm/Group | Semorinemab | Placebo | Semorinemab (Open-label Extension)
Number analyzed (Participants) | 135 | 132 | 199
Participants | 112 | 107 | 170

6. Secondary Outcome: Serum Concentration of RO7105705 at Specified Timepoints
Time Frame: Weeks 1,3,5,9,13,25,37,49, and at treatment discontinuation (up to Week 48) for Cohort 1. Weeks 1,3,5,9,13,25,37,49,61, and at treatment discontinuation (up to Week 60) for Cohort 2.
Population: The pharmacokinetic(PK)-evaluable population included all safety-evaluable participants with at least 1 post-dose serum PK sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (µg/ml)
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 135 | 0
Microgram per milliliter (µg/ml)
  Week 1 predose: number analyzed (Participants) | 130 | 0
  Week 1 predose | NA (NA) — NA = not reportable as study drug hadn't been administered yet. |
  Week 1 postdose: number analyzed (Participants) | 129 | 0
  Week 1 postdose | 1610 (27.9) |
  Week 3 predose: number analyzed (Participants) | 127 | 0
  Week 3 predose | 546 (32.1) |
  Week 3 postdose: number analyzed (Participants) | 128 | 0
  Week 3 postdose | 1980 (32.6) |
  Week 5 predose: number analyzed (Participants) | 127 | 0
  Week 5 predose | 951 (30.4) |
  Week 5 postdose: number analyzed (Participants) | 125 | 0
  Week 5 postdose | 2260 (47.0) |
  Week 9 predose: number analyzed (Participants) | 116 | 0
  Week 9 predose | 935 (32.2) |
  Week 9 postdose: number analyzed (Participants) | 117 | 0
  Week 9 postdose | 2520 (27.2) |
  Week 13 predose: number analyzed (Participants) | 118 | 0
  Week 13 predose | 943 (32.9) |
  Week 13 postdose: number analyzed (Participants) | 114 | 0
  Week 13 postdose | 2480 (31.2) |
  Week 25 predose: number analyzed (Participants) | 110 | 0
  Week 25 predose | 996 (37.1) |
  Week 25 postdose: number analyzed (Participants) | 108 | 0
  Week 25 postdose | 2420 (37.9) |
  Week 37 predose: number analyzed (Participants) | 107 | 0
  Week 37 predose | 981 (45.4) |
  Week 37 postdose: number analyzed (Participants) | 107 | 0
  Week 37 postdose | 2430 (31.1) |
  Week 49 predose: number analyzed (Participants) | 101 | 0
  Week 49 predose | 1020 (35.2) |
  Week 49 postdose: number analyzed (Participants) | 36 | 0
  Week 49 postdose | 2650 (34.2) |
  Week 61: number analyzed (Participants) | 40 | 0
  Week 61 | 1100 (26.8) |

7. Secondary Outcome: Incidence of Anti-drug Antibodies (ADAs) During the Study Relative to the Prevalence of ADAs at Baseline
Time Frame: Weeks 1,13,25,37,49, and at treatment discontinuation (up to Week 48) for Cohort 1. Weeks 1,13,25,37,49,61, and at treatment discontinuation (up to Week 60) for Cohort 2.
Population: Participants with at least one predose and one postdose ADA assessment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 135 | 132
Participants
  Baseline (BL) - positive sample: number analyzed (Participants) | 133 | 129
  Baseline (BL) - positive sample | 0 | 1
  BL - negative sample: number analyzed (Participants) | 133 | 129
  BL - negative sample | 133 | 128
  Post-BL - positive treatment emergent ADA: number analyzed (Participants) | 128 | 0
  Post-BL - positive treatment emergent ADA | 0 |
  Post-BL - negative treatment emergent ADA: number analyzed (Participants) | 128 | 0
  Post-BL - negative treatment emergent ADA | 128 |

8. Secondary Outcome: Relationship Between ADA Status and Percentage of Participants With Adverse Events
Description: Descriptive statistics will be used for assessment.
Time Frame: Up to 57 weeks for Cohort 1, and up to 69 weeks for Cohort 2.
Population: Participants with at least one predose and one postdose ADA assessment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 135 | 132
Participants | NA — Since there were no participants with ADAs, this relationship is not possible to establish. | NA — Since there were no participants with ADAs, this relationship is not possible to establish.

9. Secondary Outcome: Relationship Between ADA Status and Change From Baseline to Last Visit of Double-Blind Treatment Period in Cognitive Function as Measured by the Alzheimer's Disease Assessment Scale, Cognitive Subscale, 11-Item Version (ADAS-Cog11)
Description: Descriptive statistics will be used for assessment.
  A 70-point scale used to quantify the areas of cognitive function most often affected in Alzheimer's disease. Lower scores indicate better cognitive function.
Time Frame: Baseline to Week 49 for Cohorts 1 and 2, and Baseline to Week 61 for Cohort 2
Population: Participants with at least one predose and one postdose ADA assessment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 135 | 132
Participants | NA — Since there were no participants with ADAs, this relationship is not possible to establish. | NA — Since there were no participants with ADAs, this relationship is not possible to establish.

10. Secondary Outcome: Relationship Between ADA Status and Change From Baseline to Last Visit of Double-Blind Treatment Period in Functional Capacities as Measured by the Alzheimer's Disease Cooperative Study-Daily Living Inventory (ADCS-ADL)
Description: Descriptive statistics will be used for assessment.
  A scale used to quantify performance of activities of daily living. Scores on the ADCS-ADL range from 0-78, with higher scores indicating better ADL function.
Time Frame: Baseline to Week 49 for Cohorts 1 and 2, and Baseline to Week 61 for Cohort 2
Population: Participants with at least one predose and one postdose ADA assessment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 135 | 132
Participants | NA — Since there were no participants with ADAs, this relationship is not possible to establish. | NA — Since there were no participants with ADAs, this relationship is not possible to establish.

11. Secondary Outcome: Relationship Between ADA Status and Change From Baseline to Last Visit of Double-Blind Treatment Period on the Clinical Dementia Rating-Sum of Boxes (CDR-SB)
Description: Descriptive statistics will be used for assessment.
  A scale used to quantify the severity of symptoms of dementia. The CDR-SB is obtained through interviews of patients and informants, and disease severity is rated in 6 domains of functioning: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a 5-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). The CDR-SOB score is obtained by summing each of the domain box scores, with scores ranging from 0 to 18, with the higher values representing more severe impairment.
Time Frame: Baseline to Week 49 for Cohorts 1 and 2, and Baseline to Week 61 for Cohort 2
Population: Participants with at least one predose and one postdose ADA assessment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 135 | 132
Participants | NA — Since there were no participants with ADAs, this relationship is not possible to establish. | NA — Since there were no participants with ADAs, this relationship is not possible to establish.

12. Secondary Outcome: Relationship Between ADA Status and Change From Baseline to Last Visit of Double-Blind Treatment Period on the Mini-Mental State Examination (MMSE)
Description: Descriptive statistics will be used for assessment.
  The Mini Mental State Examination (MMSE) is a brief clinical cognitive examination commonly used to screen for dementia and other cognitive deficits that has a total score of 0-30. Higher scores indicate better cognitive function.
Time Frame: Baseline to Week 49 for Cohorts 1 and 2, and Baseline to Week 61 for Cohort 2
Population: Participants with at least one predose and one postdose ADA assessment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 135 | 132
Participants | NA — Since there were no participants with ADAs, this relationship is not possible to establish. | NA — Since there were no participants with ADAs, this relationship is not possible to establish.

13. Secondary Outcome: Relationship Between ADA Status and Serum Concentration of RO7105705 at Specified Timepoints
Description: Descriptive statistics will be used for assessment.
Time Frame: as for outcome 7
Population: Participants with at least one predose and one postdose ADA assessment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 135 | 132
Participants | NA — Since there were no participants with ADAs, this relationship is not possible to establish. | NA — Since there were no participants with ADAs, this relationship is not possible to establish.

14. Secondary Outcome: Relationship Between ADA Status and Incidence of Anti-Drug Antibodies (ADAs) During the Study Relative to the Prevalence of ADAs at Baseline
Description: Descriptive statistics will be used for assessment.
Time Frame: as for outcome 7
Population: Participants with at least one predose and one postdose ADA assessment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Semorinemab | Placebo
Number analyzed (Participants) | 135 | 132
Participants
  Positive Sample at BL | 0 | 1
  Positive Sample post BL | NA — Since there were no participants with ADAs, this relationship is not possible to establish. | NA — Since there were no participants with ADAs, this relationship is not possible to establish.

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (approximately 4 years and 7 months)
Description: The safety population included all randomized participants who received at least one dose of either semorinemab or placebo.
Groups:
- Semorinemab (Double Blind): Semorinemab was administered intravenously in the double-blind treatment period
- Semorinemab (OLE): Semorinemab was administered intravenously in the optional open-label extension period.
Arm/Group | Semorinemab (Double Blind) | Placebo | Semorinemab (OLE)
All-Cause Mortality (participants affected / at risk) | 1/135 | 3/132 | 2/199
Serious Adverse Events (participants affected / at risk) | 23/135 | 22/132 | 37/199
Other Adverse Events (participants affected / at risk) | 78/135 | 74/132 | 122/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semorinemab (Double Blind) (N=135) | Placebo (N=132) | Semorinemab (OLE) (N=199)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 4 (4)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Upper motor neurone lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 3 (3) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary fistula (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (5)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semorinemab (Double Blind) (N=135) | Placebo (N=132) | Semorinemab (OLE) (N=199)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 5 (6) | 10 (10)
Nasopharyngitis (Infections and infestations) | 9 (10) | 3 (3) | 5 (5)
Urinary tract infection (Infections and infestations) | 11 (14) | 16 (19) | 27 (36)
Fall (Injury, poisoning and procedural complications) | 14 (20) | 19 (28) | 37 (64)
Infusion related reaction (Injury, poisoning and procedural complications) | 14 (30) | 5 (9) | 14 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4) | 11 (12)
Dizziness (Nervous system disorders) | 8 (8) | 9 (11) | 7 (8)
Headache (Nervous system disorders) | 11 (14) | 9 (10) | 10 (13)
Agitation (Psychiatric disorders) | 8 (8) | 8 (8) | 18 (19)
Anxiety (Psychiatric disorders) | 9 (11) | 12 (12) | 11 (11)
Depression (Psychiatric disorders) | 10 (11) | 7 (7) | 6 (6)
Insomnia (Psychiatric disorders) | 7 (7) | 3 (3) | 13 (13)
Hypertension (Vascular disorders) | 8 (10) | 5 (5) | 5 (5)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT03828747/Prot_SAP_000.pdf